CLINICAL TRIAL: NCT01932736
Title: Functional Manifestations of Pressure Changes in the Middle Ear System: An fMRI Study
Brief Title: Functional Manifestations of Pressure Changes in the Middle Ear System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, J. Douglas Swarts, Research Associate Professor of Otolaryngology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO13030623
Record Dates: First submitted 2013-08-09; First posted 2013-08-30 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Middle-ear Function
Keywords: middle ear; Eustachian tube; fMRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy volunteers (Experimental): healthy volunteers undergo pressure changes in ear canal
  Interventions: Other: changing ear canal pressure

INTERVENTIONS:
Other: changing ear canal pressure — ear canal pressure changes: pressure varied from +/-40 decapascals

SUMMARY:
This study is looking at whether functional magnetic resonance imaging (fMRI) can see if and when the brain responds to pressure stimulations of the eardrum. The study requires 2 visits, 1 for screening to determine eligibility and 1 for the fMRI. This study will help to understand how the middle ear system is controlled, which may have an impact on how people with middle ear disease are treated.

DETAILED DESCRIPTION:
Otitis media is a ubiquitous disease in young children which can persist through adolescence, and arise or recur in adults. A consequence of an infection and/or Eustachian tube dysfunction, it manifests as an effusion that disrupts the normal impedance matching function of tympanic membrane-ossicular chain system. Eustachian tube dysfunction prevents the equilibration of middle ear pressures and drainage of the accumulated effusion. It is thought that middle ear status modulates the function of the Eustachian tube via afferent signals processed centrally resulting in changes in its tonus or muscular function. This pilot study of right-handed 21-35 year olds of either sex will validate a published fMRI method for visualizing cortical brain activation in response to external ear canal pressure changes (N=5). The outcome measure is intensity changes of the cortex associated with applied stimuli.

ELIGIBILITY:
Inclusion Criteria:

* 21-35 years of age
* right-handed

Exclusion Criteria:

* left-handedness or ambidexterity
* fMRI safety reasons (ferromagnetic material in their bodies, epilepsy, claustrophobia
* history of middle ear/tympanic membrane surgery (tympanostomy tubes)
* abnormal otoscopic findings and/or tympanometry on physical exam
* pregnancy

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
changes in brain activation during pressure changes | 1 hour (Visit 2, during fMRI)
  Subjects will have fMRIs while pressure is varied in the right ear (+/-40 decapascals). Changes in brain activation during pressure changes will be measured by fMRI during approximately 1 hour scanning time.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Swarts, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Middle Ear Physiology Laboratory, University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No